CLINICAL TRIAL: NCT01456767
Title: The Effects of Oral Administration of Lactobacillus Plantarum WCFS1, Lactobacillus Plantarum CIP104448, and Lactobacillus Plantarum CIP104450 on Small Intestinal Mucosa and Barrier Function
Brief Title: Effects of Administration of L.Plantarum WCFS1, L.Plantarum CIP104448, L.Plantarum CIP104450 on Small Intestinal Mucosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: NL35728.068.11/METC11-2-011
Record Dates: First submitted 2011-10-10; First posted 2011-10-21 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Gastro Intestinal Infection
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lactobacillus plantarum WCFS1 (Active Comparator): Al study subjects will in randomized sequence participate in this arm (7-days supplementation period of Lactobacillus plantarum WCFS1).
  Each arm represents a 7-days supplementation period (with probiotics or placebo). The 7-days supplementation period will be followed by a month washout time after which the next supplementation period with another probiotic (or placebo) will start. The sequence is randomized and double blind. The different measurements will be performed at baseline and after each supplementation period.
  Interventions: Dietary Supplement: Probiotics
- Lactobacillus plantarum CIP104448 (Active Comparator): Al study subjects will in randomized sequence participate in this arm (7-days supplementation period of Lactobacillus plantarum CIP104448).
  Each arm represents a 7-days supplementation period (with probiotics or placebo). The 7-days supplementation period will be followed by a month washout time after which the next supplementation period with another probiotic (or placebo) will start. The sequence is randomized and double blind. The different measurements will be performed at baseline and after each supplementation period.
  Interventions: Dietary Supplement: Probiotics
- Lactobacillus plantarum CIP104450 (Active Comparator): Al study subjects will in randomized sequence participate in this arm (7-days supplementation period of Lactobacillus plantarum CIP104450).
  Each arm represents a 7-days supplementation period (with probiotics or placebo). The 7-days supplementation period will be followed by a month washout time after which the next supplementation period with another probiotic (or placebo) will start. The sequence is randomized and double blind. The different measurements will be performed at baseline and after each supplementation period.
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): Al study subjects will in randomized sequence participate in this arm (7-days supplementation period of a placebo).
  Each arm represents a 7-days supplementation period (with probiotics or placebo). The 7-days supplementation period will be followed by a month washout time after which the next supplementation period with another probiotic (or placebo) will start. The sequence is randomized and double blind. The different measurements will be performed at baseline and after each supplementation period.
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — Bacterial supplements (Lactobacillus plantarum WCFS1, Lactobacillus plantarum CIP104448, and Lactobacillus plantarum CIP104450) will be prepared in the food-grade pilot plant of NIZO food research. Exactly 1x10^11 life bacteria are consumed by each participant.
  Consumption of this amount of life bacteria is in line with earlier human studies and routinely reached by the consumption of dairy. As a placebo, the same drink will be used without addition of bacterial cells.

SUMMARY:
The design of this study conforms to a randomized double-blind placebo-controlled cross-over design.

The objective of the study is to assess the effect of three probiotics (Lactobacillus plantarum WCFS1, Lactobacillus plantarum CIP104448, and Lactobacillus plantarum CIP104450) on intestinal epithelial permeability and the immune system, in at least 8 healthy subject.

The effect of the three different probiotics and a placebo will be assessed on every subject in random sequence.

Prior to the start of a 7-days supplementation period (one of the three probiotic supplements or placebo), blood samples will be obtained and small intestinal permeability will be assessed by measuring the urinary extraction ratios of ingested water-soluble, non-degradable test probes, with and without indomethacin challenge (to compromise the gut). After each supplementation period the gut will be stressed again by the indomethacin protocol, followed by measurement of small intestinal permeability, whereupon blood samples will be taken and duodenal tissue samples will be obtained by standard gastroduodenoscopy. Each supplementation period will start 1 month after finishing the pervious test episode, in randomized sequence.

The primary objective of this study is to assess the effects of Lactobacillus plantarum WCFS1, Lactobacillus plantarum CIP104448, and Lactobacillus plantarum CIP104450 on intestinal epithelial permeability. Secondary objectives are to assess the effects on immune modulation, gene expression of peripheral blood mononuclear cells, small intestine epithelial gene regulation and tight junction proteins modulation, infiltration of immune cells in intestinal mucosa and immune markers in blood plasma.

The investigators hypothesize that Lactobacillus plantarum WCFS1, Lactobacillus plantarum CIP104448, and Lactobacillus plantarum CIP104450 will, each separately, significantly affect the innate immune system and intestinal permeability in humans.

ELIGIBILITY:
Inclusion Criteria:

* Based on medical history and previous self-admitted examination, no gastrointestinal complaints can be defined.
* Age between 18 and 65 years.
* BMI between 20 and 30 kg/m2.

Exclusion Criteria:

* History of severe cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological diseases, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol.
* Use of medication, including vitamin supplementation, except oral contraceptives, within 14 days prior to testing.
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 180 days prior to the study.
* Major abdominal surgery interfering with gastrointestinal function (uncomplicated appendectomy, cholecystectomy and hysterectomy allowed, and other surgery upon judgement of the principle investigator).
* Pregnancy, lactation.
* Excessive alcohol consumption (>20 alcoholic consumptions per week).
* Smoking.
* Blood donation within 3 months before or after the study period.
* Self-admitted HIV-positive state.
* Known hypersensitivity or history of allergic reactions towards intake of non-steroidal anti-inflammatory drugs (NSAIDs) or non- or low caloric sweeteners of any kind.
* History of any side effects towards intake of pro- or prebiotic supplements of any kind.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in sugar recovery in urine, as indicator of intestinal permeability, after seven days probiotics supplementation. | Permeability will be assessed at baseline (3 days before supplementation), at baseline after indomethacin administration (1 day before supplementation) and after the 7-days probiotics supplementation period (again after indomethacin administration).
  The barrier function test is based on a comparison of intestinal permeation of a larger molecule with that of a smaller molecule. The subject will ingest a sugar drink containing sucrose, lactulose, L-rhamnose, sucralose and erythritol after an overnight fast. All sugar probes are accepted and validated parameters of integrity of the intestinal barrier, and proved an accurate estimation of mucosal damage.
  Urine samples will be obtained to measure sugar recovery. The sugar molecules will be determined by fluorescent detection high-pressure liquid chromatography (HPLC).

SECONDARY OUTCOMES:
Differences of measurements in duodenal biopsy specimens between the separate arms. | Duodenal biopsy specimens will be obtained at the end of each probiotics supplementation period (one day after the seven day supplementation).
  * Tight junction proteins with immunofluorescent labelling and PCR quantification of perijunctional actin, myosin, ZO-1, claudin-3, occludin, myosin light chain kinase, and phosphorylated myosin light chain
  * Transcriptomics: Affymetrix genome-wide microarrays, Validation and semi-quantification of selected genes by qPCR
  * Markers of immune activation: Infiltration of immune cells by immunofluorescent staining
  * Biochemical analysis of myeloperoxidase (MPO)
Change in measurements in whole blood, after the seven days probiotics supplementation period. | Measurements in whole blood will be carried out at baseline (3 days before supplementation) and after the 7-days probiotics supplementation period.
  * Quantify immune cell populations (T helper cells, cytotoxic T cells, CD25+ effector T cells, CD69+ effector T cells, regulatory T cells, and NK-cells)
  * Biomarkers of immune stimulation (the human cytokines IL-10, TGF-β, IL-12p40 subunit, IL-12p70 subunit, IL-1β, IL-2, IL-6, IL-4, IL-17, IL-22 and IFN-γ, TNFα)
  * Transcriptomics on peripheral blood mononuclear cells: affymetrix genome-wide microarrays, validation and semi-quantification of selected genes by qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Ad Masclee, Prof. dr., Principal Investigator — Maastricht University Medical Center; Freddy Troost, Dr., Principal Investigator — Maastricht University Medical Center; Zlatan Mujagic, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Health, Medicine and Life Sciences, Maastricht, Limburg, Netherlands